CLINICAL TRIAL: NCT01695759
Title: Evaluation of Clinical Efficacy and Immunogenicity of Drug Eritromax® at Blau Farmacêutica S.A. Compared to Eprex®, Produced by Janssen-Cilag Laboratory in Participants With Secondary Anemia to Chronic Kidney Disease.
Brief Title: Clinical Efficacy of Two Erythropoietin Drug in Participants With Secondary Anemia to Chronic Kidney Disease.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Collaborators: Blau Farmaceutica S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EPOBLA1011; Emenda 04 - 11/May/2015 (Other: Azidus Brasil Pesquisa Científica e Desenvolvimento Ltda.)
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Chronic Kidney Disease; Anemia
Keywords: Anemia Secondary; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia | interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epoetin alpha (Experimental): Participants assigned to this arm will receive two subcutaneous administrations per week of 50 UI/kg of Epoetin alpha (Eritromax), totaling 100 UI/kg/week. After the first four weeks of treatment, once a month throughout the study the medication dose can be adjusted by the study Investigator according to the laboratory results.
  Interventions: Drug: Epoetin alpha
- Eprex (Active Comparator): Participants assigned to this arm will receive two subcutaneous administrations per week of 50 UI/kg of Epoetin alpha (Eprex), totaling 100 UI/kg/week. After the first four weeks of treatment, once a month throughout the study the medication dose can be adjusted by the study Investigator according to the laboratory results.
  Interventions: Drug: Eprex

INTERVENTIONS:
Drug: Epoetin alpha — Participants assigned to this arm will receive two subcutaneous administrations per week of 50 UI/kg of Epoetin alpha (Eritromax), totaling 100 UI/kg/week. After the first four weeks of treatment, once a month throughout the study the medication dose can be adjusted by the study Investigator according to the laboratory results.
  Arms: Epoetin alpha
Drug: Eprex — Participants assigned to this arm will receive two subcutaneous administrations per week of 50 UI/kg of Epoetin alpha (Eprex), totaling 100 UI/kg/week. After the first four weeks of treatment, once a month throughout the study the medication dose can be adjusted by the study Investigator according to the laboratory results.
  Other Names: Epoetin alpha
  Arms: Eprex

SUMMARY:
This is a prospective, randomized, multicenter, parallel, placebo-controlled, phase III study for evaluation of clinical efficacy and immunogenicity of drug Eritromax® - (rHuEPO Blau Farmacêutica S/A.) compared to Eprex® (Janssen-Cilag rHuEPO) for the treatment of patients with secondary anemia to chronic kidney disease (CKD), throughout the correction phase by assessing the change in hemoglobin levels.

DETAILED DESCRIPTION:
This is a phase III study, in which participants with secondary anemia to chronic kidney disease will receive two subcutaneous injection of 50 UI/Kg of the investigational product (Eritromax®) or Eprex® per week. After four weeks of treatment, the dose of drugs will be change by clinical judged throughout study according to laboratory results. The evidence of efficacy will be evaluated by hemoglobin levels alteration throughout the correction phase (first four weeks). Secondary efficacy and safety endpoints will be assessed by: maintenance of hemoglobin levels (baseline vs. end of treatment) over maintenance phase; dose of EPO required during correction and maintenance phase; Transfusion needs; report of adverse events (including type, frequency, intensity, serioussness, severity and relation to the investigation product) throughouht 12 months of follow-up. Additionally, the immunological response of products over study will be evaluated by quantification of anti-erythropoietin every six months.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and agree to all the purposes of the study by signing and dating ICF;
2. Male or female participantes, regardless of race or social class;
3. Participants aged ≥18 and ≤70 years;
4. Bearer dialysis-dependent CKD (hemodialysis and peritoneal dialysis *);
5. Clinical diagnosis of anemia, characterized as hemoglobin levels <10g/dL before the start of the study;
6. Adequate dialysis: Kt / V ≥ 1.2 for hemodialysis patients (based on the calculation of Daugirdas II) and ≥ 1.7 for patients on peritoneal dialysis;
7. Adequate iron stores (TSAT> 20% and serum ferritin> 100ng/ml) prior to initiation of treatment with erythropoietin.

Exclusion Criteria:

1. Participation in clinical trials in the 12 months preceding the survey;
2. Patients with uncontrolled hypertension, with mean above 180/100mmHg and whose requiring hospitalization in the last 6 months;
3. Presence of other causes of anemia than CKD, such as bleeding, hemolysis, pernicious anemia and hemoglobinopathies;
4. Patients who present changes or clinical abnormalities, qualified as interfering changes, such as severe hyperparathyroidism (iPTH> 1000 pg / mL), severe congestive heart failure (NYHA Class IV), acute myocardial infarction within the last 3 months, or active neoplasia in follow-up, severe liver disease, active infection (leukocyte changes), history of aluminum toxicity or scheduled surgery, pregnancy or lactation;
5. Patients who have a known hypersensitivity to any component of the formulation and to products derived from mammalian cells;
6. Prior therapies with erythropoietin for less than 3 months;
7. Realization transfusion for less than 3 months;
8. Any situation at the discretion of the Principal Investigator interfere with study data.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change of hemoglobin levels at correction phase (baseline vs end of treatment) | until 6 months
  In the correction phase, change in serum Hb levels (baseline vs. end of initial treatment (EOIT) = levels of Hb presented before the V0 treatment compared to the Hb levels presented at the end of the correction phase) will be evaluated for a maximum period of 6 months after starting treatment. This one parameter will be demonstrated through: Percentage of participants achieving Hb levels within the target (≥ 10.5 to ≤ 12 g / dL).

SECONDARY OUTCOMES:
Maintenance of hemoglobin levels | until the end of 12 months
  Will be evaluated by porcentage of participants whose Hb levels remained within the therapeutic range (≥10,5 a ≤ 12 g/dL).
Adjustment of EPO dose required during correction and/or maintenance phase | until the end of 12 months
  Will be evaluated by mean dose of EPO used between groups and number of participants that needed of dose adjustment over correction and/or maintenance phase.
Transfusion needs | until the end of 12 months
  Will be evaluated by porcentage of participants that needed of blood transfusion throughout the study.
Report of Adverse Events | until the end of 12 months
  Will be evaluated by report of adverse events throughout the study. The Adverse events will be classified about the type, frequency, intensity, seriousness, severity and relation to the investigational product.

OTHER OUTCOMES:
Immunological Response | every six months
  The immunological response induced by epoetin alpha will be evaluated by quantification of anti-erithropoetin antibodies, every six months.

CONTACTS AND LOCATIONS:
Overall Officials: Regiane Braga, Analyst, Study Chair — Blau Farmaceutica S.A.
Locations (10):
- Brazil (10):
  - Clínica Senhor do Bomfim Ltda, Feira de Santana, Estado de Bahia
  - Instituto Scribner de Ensino, Pesquisa, Ciência e Tecnologia, Curitiba, Paraná
  - Fundação Universitária de Caxias do Sul - Instituto de Pesquisa Clínica para Estudos Multicêntricos, Caxias do Sul, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - União Brasileira de Educação e Assistência Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Fundação Pró-Rim, Joinville, Santa Catarina
  - Hospital de Ensino Padre Anchieta, São Bernardo do Campo, São Paulo
  - CMIN - Clínica De Medicina Interna E Nefrologia, São Paulo
  - Fundação Oswaldo Cruz (Hospital do Rim e Hipertensão), São Paulo
  - Real e Benemérita Associação Portuguesa de Beneficência São Paulo (Hospital Beneficência Portuguesa), São Paulo

IPD SHARING:
Plan to Share IPD: Undecided